CLINICAL TRIAL: NCT01355926
Title: Flexible Fiber-based CO2 Laser Versus Monopolar Cautery for Resection of Benign, Pre-malignant And Malignant Oral Cavity Lesions: A Single Center Randomized Controlled Trial Assessing Pain and Quality of Life Following Surgery
Brief Title: A Single Center Randomized Controlled Trial Assessing Pain and Quality of Life Following Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: OMNIGUIDE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-034
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Head and Neck Cancer
Keywords: Flexible Fiber-based CO2 Laser; Monopolar Cautery; Oral Cavity Lesions; Quality of life; Assessing Pain; 11-034
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Flexible Fiber-based CO2 Laser (Experimental): In the CO2 excised group, the resection will be performed at 15W, at a distance of 1cm from the tissue. Here too, if required, the bipolar will be used to achieve hemostasis The study will focus on post operative pain and quality of life outcomes for both surgical interventions.
  Interventions: Other: Flexible Fiber-based CO2 Laser, Quality of Life forms
- electrocautery resection (Experimental): In the electrocautery excised group, the cut and coagulation modes used will be each at 25 Malis power setting. First, cut mode will be used to mark out the lesion. Subsequently, coagulation mode will be used for excision. Bipolar cautery will then be used at 25 Malis for hemostasis. The study will focus on post operative pain and quality of life outcomes for both surgical interventions.
  Interventions: Other: electrocautery resection and quality of life forms

INTERVENTIONS:
Other: Flexible Fiber-based CO2 Laser, Quality of Life forms — . Post operative pain will be measured pre-operatively, and post-operatively on post-operative day (POD) 1, 3, 7, 14, 21 and 28 using a numerical pain rating scale. The secondary outcomes will be measured pre-operatively and post-operatively using the University of Washington Quality of Life questionnaire specific for head and neck version 4 (UW-QOL version 4) and the Performance Status Scale for head and neck cancer (PPS-HN) on days 7, 14 and 28. Other secondary aims will be measured intra-operatively and time to return to work and time to normal diet will be measured during timeframes of POD 1, 3, 7,14, 21 and 28.
  Arms: Flexible Fiber-based CO2 Laser
Other: electrocautery resection and quality of life forms — Post operative pain will be measured pre-operatively, and post-operatively on post-operative day (POD) 1, 3, 7, 14, 21 and 28 using a numerical pain rating scale. The secondary outcomes will be measured pre-operatively and post-operatively using the University of Washington Quality of Life questionnaire specific for head and neck version 4 (UW-QOL version 4) and the Performance Status Scale for head and neck cancer (PPS-HN) on days 7, 14 and 28. Other secondary aims will be measured intra-operatively and time to return to work and time to normal diet will be measured during timeframes of POD 1, 3, 7,14, 21 and 28.
  Arms: electrocautery resection

SUMMARY:
The purpose of this study is to help us to better understand the effects of two different types of surgical techniques on pain and quality of life in patients with precancerous lesions or early stage mouth cancers.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven diagnosis or clinical diagnosis of any benign oral cavity lesion. Pre-surgical biopsy will not be required if lesion is suspected to be benign.
* Biopsy proven diagnosis or clinical diagnosis of premalignant oral cavity lesions (leukoplakia, erythroplakia, lichen planus, dysplasia)Pre-surgical biopsy will not be required if lesion is suspected to be benign.
* Biopsy proven diagnosis of small superficial oral cavity SCC (stage T1N0) requiring resection without the need for neck dissection.
* All pathology will be reviewed at MSK to confirm diagnosis.
* The lesion plus the resection margin should not exceed 4.0 cm circumferentially.
* Planned to undergo surgical treatment by resection without flap reconstruction and without neck dissection.
* All patients age 18 years of age and older.
* Karnofsky performance score over 60.

Patients on blood thinners (aspirin or Coumadin) will be asked to stop medications 7 days prior to surgery. In the case of Coumadin, patients are switched to lovenox 7 days prior to surgery and this is stopped the day before surgery. Following surgery aspirin or Coumadin are recommenced 48 hours postop.

Exclusion Criteria:

* Patients with previous Head and Neck radiation
* Pregnant or lactating female patients.
* Patients with oral cavity squamous cell cancer requiring neck dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
To demonstrate that for treatment of oral benign, oral leukoplakia and superficial T1N0M0 oral cavity lesions, CO2-fiber based resection generates less thermal damage compared to monopolar cautery | 1 month
  Leading to improved patient quality of life and post-operative recovery as manifested by reduced post-operative pain. Post operative pain will be measured pre-operatively, and post-operatively on post-operative day (POD) 1, 3, 7, 14, 21 and 28 using a numerical pain rating scale.

SECONDARY OUTCOMES:
to evaluate differences between the two surgical modalities | 1 month
  in terms of intra-operative parameters, postoperative quality of life and cost effectiveness will be measured intra-operatively and time to return to work and time to normal diet will be measured during timeframes of POD 1, 3, 7,14, 21 and 28.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Ganly, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm